CLINICAL TRIAL: NCT04964024
Title: SaRS-Cov-2 Antibodies Following Exposure to COVID-19 and/or Vaccination in Nursing Homes
Brief Title: SaRS-Cov-2 Antibodies Following Exposure to Coronavirus Disease 2019 (COVID-19) and/or Vaccination in Nursing Homes
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pr Athanase BENETOS, Athanase Benetos, Clinical Professor, Head of the Dpt of Geriatrics, Central Hospital, Nancy, France
Other Study IDs: EHPAD-COVID-19
Record Dates: First submitted 2021-06-26; First posted 2021-07-15 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: COVID-19 Infection
Keywords: SARS-CoV-2; Antibodies; Vaccination; Nursing Homes
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Residents in Nursing homes
  Interventions: Diagnostic Test: SARS-CoV-2 antibodies
- Health professionals in Nursing homes
  Interventions: Diagnostic Test: SARS-CoV-2 antibodies

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 antibodies — Analysis of the results of the serological response to COVID-19 and/or Vaccine

SUMMARY:
Presence of SaRS-Cov-2 antibodies following exposure to Coronavirus Disease 2019 (COVID-19) and/or vaccination is a major indicator of immunization. Few data exit about serology response in nursing homes (NHs), i.e. in the most vulnerable population for developing severe forms of the disease.

Residents and health professionals in 9 nursing homes (NHs) with SaRS-Cov-2 antibodies detection after exposure (either COVID-19 or vaccine) All biological tests were performed in the frame of the standard care of residents and health professionals and all participants did not express opposition for using anonymously their data for the purpose of this academic analysis. In addition all Directors and Physicians of these NHs accepted to participate in this study

ELIGIBILITY:
Inclusion Criteria:

For Residents:

* Living in one of the 9 Nursing Homes that participate in this study
* Having a SARS-COV-2 post vaccination serology.
* Having no objection for using the results of the serology for the purpose of this analysis

For Health Professionals:

* Working in one of the 9 Nursing Homes that participate in this study,
* Having a SARS-COV-2 post vaccination serology.
* Having no objection for using the results of the serology for the purpose of this analysis

Exclusion Criteria:

* None

Ages: 20 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of the 9 Nursing Homes that participate in this study Health professionals working these Nursing Homes
Sampling Method: Non-Probability Sample
Enrollment: 1293 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Levels of SARS-COV-2 antibodies | Through study completion average 6 months Retrospective analysis
  Study of the SARS-COV-2 antibodies according to the history of COVID-19 and vaccinal status in Nursing Home residents and in health professionals

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Université de Lorraine, Vandœuvre-lès-Nancy, US and Canada Only, France

IPD SHARING:
Plan to Share IPD: Undecided
The database can be used by other groups but only for academic purposes